CLINICAL TRIAL: NCT06917898
Title: Fentanyl Versus Midazolam During Spinal Block With Bupivacaine for Elective Cesarean Delivery: a Prospective Randomized Double-blind Clinical Trial.
Brief Title: Fentanyl Versus Midazolam as an Adjunct to Spinal Anesthesia
Acronym: Spinal Block
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Omar Rajab, Chairman of Anesthesia Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MGH-07-24001
Record Dates: First submitted 2025-04-07; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy Female Volunteer
Keywords: Fentanyl; Midazolam; Obstetrical Anesthesia; Cesarean Section; Bupivacaine; Spinal Anesthesia
MeSH Terms: interventions — Anesthesia, Spinal; Bupivacaine; Fentanyl; Midazolam

STUDY DESIGN:
Intervention Model Description: The study design implemented will be a Double-blinded, prospective randomized clinical trial at Makassed General Hospital comparing two groups, Group (M) for midazolam and Group (F) for fentanyl where both patients and physicians will be unaware (blinded) of which drug was used during the spinal neuraxial block. Patients aged 18-45 with American Society of Anesthesia (ASA) class II will be included in the study.
  Patients excluded from the clinical trial include those with contraindications to spinal anesthesia such as infection at injection site, bleeding coagulopathies with risk of spinal hematoma formation, and history of allergies to bupivacaine, opioids, or midazolam. Exclusion criteria also included patients with history of opioid substance abuse, pre-eclampsia or eclampsia, uncontrolled diabetes mellitus, and significant cardiac, renal, and hepatic morbidity (i.e., ASA class III patients).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Fentanyl (Active Comparator)
  Interventions: Drug: Spinal Anesthesia with Bupivacaine and Fentanyl
- Intrathecal Midazolam (Active Comparator)
  Interventions: Drug: Spinal Anesthesia with Bupivacaine and Midazolam

INTERVENTIONS:
Drug: Spinal Anesthesia with Bupivacaine and Fentanyl — 25 mcg Fentanyl 12.5 mg Bupivacaine
  Arms: Intrathecal Fentanyl
Drug: Spinal Anesthesia with Bupivacaine and Midazolam — 2 Mg Midazolam 12.5 mg Bupivacaine
  Arms: Intrathecal Midazolam

SUMMARY:
It is well documented in the practice of anesthesia the effectiveness of bupivacaine when added with other adjuvants including midazolam, opioids, and ketamine during neuraxial spinal block for cesarean delivery, however comparison of the superiority of midazolam 2mg over fentanyl 25 micrograms or vice versa with bupivacaine during cesarean delivery has not been established and if performed diligently, could potentially change our understanding and current practice for better patient outcomes.

DETAILED DESCRIPTION:
A study published on Jan - Feb 2024 has compared adjuvants fentanyl 25 micrograms and midazolam 2mg when added to Levobupivacaine for patients undergoing cesarean section with Midazolam being the superior drug of choice with less side effects. [1] Another study done around our locality at the American University of Beirut compared the postoperative analgesic effect of ketamine and fentanyl when added to bupivacaine in patients undergoing cesarean section with results conclusive of equally effective post cesarean pain control. [2] One study compared intrathecal midazolam 2mg with intrathecal fentanyl 12.5 micrograms with bupivacaine [3], and results elucidated equal surgical analgesia during the operation in contrast to the superior Midazolam 2mg vs the intrathecal fentanyl 25 micrograms when added to levobupivacaine mentioned in the first study. Current literature is void of studies comparing intrathecal fentanyl 25 micrograms vs intrathecal midazolam 2mg when added to bupivacaine for cesarean delivery.

Study objectives:

Comparative studies are available for different adjuvants when administered along with bupivacaine or levobupivacaine, but the specific aim and target of this study is to compare Hyperbaric Bupivacaine 0.5% 12.5 mg with fentanyl 25 micrograms (2 ml) versus Hyperbaric Bupivacaine 0.5% 12.5 mg with midazolam 2mg (2 ml) for cesarean delivery.

Levobupivacaine is not as readily available as bupivacaine in our population. Opioids have significantly more side effects when administered intrathecally including pruritus, respiratory depression, post operatively nausea and vomiting, and any attempt to decrease their usage to improve patient satisfaction without compromising the overall analgesic effect should be pursued. The results from this study could potentially change current practice in our hospital and across local and national areas respectively.

This study aims to provide conclusive data about the superiority of midazolam in reduction of postoperative pain, reduction of postoperative rescue analgesia, the quality of sensory block, and the reduction in side effects when administered with Bupivacaine as opposed to Levobupivacaine which was demonstrated in the study [1] mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-45 with American Society of Anesthesia (ASA) class II will be included in the study.

Exclusion Criteria:

* patients with history of opioid substance abuse
* pre-eclampsia or eclampsia
* Gestational Hypertension
* uncontrolled diabetes mellitus
* significant cardiac, renal, and hepatic morbidity (i.e., ASA class III patients).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant female participants
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
rescue analgesia | 24 Hours
  The primary outcome is the timing of the first analgesia requested postoperatively (i.e., the rescue analgesia).

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khezri MB, Tahaei E, Atlasbaf AH. COMPARISON OF POSTOPERATIVE ANALGESIC EFFECT OF INTRATHECAL KETAMINE AND FENTANYL ADDED TO BUPIVACAINE IN PATIENTS UNDERGOING CESAREAN SECTION: A PROSPECTIVE RANDOMIZED DOUBLE-BLIND STUDY. Middle East J Anaesthesiol. 2016 Feb;23(4):427-36. PMID 27382812
- [Background] Abdelrady MM, Fathy GM, Abdallah MAM, Ali WN. Comparison of the effect of adding midazolam versus fentanyl to intrathecal levobupivacaine in patients undergoing cesarean section: double-blind, randomized clinical trial. Braz J Anesthesiol. 2024 Jan-Feb;74(1):744385. doi: 10.1016/j.bjane.2022.06.001. Epub 2022 Jun 11. PMID 35700752
- See also: Related Info — https://www.jebmh.com/abstract/comparison-of-intrathecal-fentanyl-and-midazolam-as-an-adjuvant-to-bupivacaine-for-enhancing-the-quality-of-subarachnoid-82103.html